CLINICAL TRIAL: NCT02335853
Title: Association Between Metabolic Syndrome and Serum Nerve Growth Factor Levels in Women With Overactive Bladder
Acronym: NGF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014/11/02
Record Dates: First submitted 2015-01-02; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Overactive Bladder
Keywords: urinary bladder; nerve growth factor; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- women with metabolic syndrome and overactive bladder: women with urinary urgency+frequency+nocturia and current ATP III criteria define the metabolic syndrome as the presence of any three of the following five traits:
  1. Abdominal obesity, defined as a waist circumference in men ≥88 cm
  2. Serum triglycerides ≥150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides
  3. Serum HDL cholesterol <40 mg/dL (1 mmol/L) in men and <50 mg/dL (1.3 mmol/L) in women or drug treatment for low HDL-C
  4. Blood pressure ≥130/85 mmHg or drug treatment for elevated blood pressure
  5. Fasting plasma glucose (FPG) ≥100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose
- women with overactive bladder: women with urinary urgency+frequency+nocturia
- healthy control group: women not overactive bladder and metabolic syndrome

SUMMARY:
Nerve growth factor (NGF-R) receptors are between the detrusor muscle fibers and can cause afferent signals. Metabolic syndrome and obesity have been advocated to be risk factors for the development of overactive bladder.

DETAILED DESCRIPTION:
Overactive bladder is a clinical syndrome characterized urgency, frequency and nocturia. Infection or other obvious causes must be excluded. The overactive bladder is loss of inhibition of the detrusor muscle during the filling or emptying of the bladder.

Specific receptors and neurotransmitters have role in development of overactive bladder. These includes adrenergic, cholinergic, non-adrenergic, non-cholinergic receptors and interstitial cells.

Nerve growth factor (NGF-R) receptors are between the detrusor muscle fibers and can cause afferent signals. Metabolic syndrome and obesity have been advocated to be risk factors for the development of overactive bladder. The investigators believe that our findings will shed light on treatment.

ELIGIBILITY:
Inclusion Criteria:

* women with urgency, nocturia and frequency
* Abdominal obesity, defined as a waist circumference in men ≥88 cm
* Serum triglycerides ≥150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides
* Serum HDL cholesterol <40 mg/dL (1 mmol/L) in men and <50 mg/dL (1.3 mmol/L) in women or drug treatment for low HDL-C
* Blood pressure ≥130/85 mmHg or drug treatment for elevated blood pressure
* Fasting plasma glucose (FPG) ≥100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose

Exclusion Criteria:

* Chronic obstructive pulmonary disease allergy
* Psychiatric disorders
* Urinary tract infection
* Neurological diseases
* Metabolic diseases
* Pure stress or mixed urinary incontinence
* History of pelvic surgery
* Diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women with overactive bladder
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
nerve growth factor levels | 3 months
  association between nerve growth factor levels and overactive bladder

SECONDARY OUTCOMES:
urge incontinence | 3 months
  number of urge incontinence
overactive bladder symptoms | 3 months
  number of nocturia,urgency,frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)